CLINICAL TRIAL: NCT02449369
Title: Intra-Venous Acetaminophen and Muscle Relaxants After Total Knee Arthroplasty (TKA). Prospective, Randomized, Open-label Trial to Determine if Switching From Oral to Intravenous Acetaminophen and Orphenadrine for 48 Hours After TKA Improves Outcomes.
Brief Title: Intra-Venous Acetaminophen and Muscle Relaxants After Total Knee
Acronym: IVAM
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: AdventHealth (Other)
Collaborators: Sagent Pharmaceuticals Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 521770
Record Dates: First submitted 2015-05-14; First posted 2015-05-20 (Estimated); Last update posted 2017-08-31 (Actual); Status verified 2017-08

CONDITIONS: Unilateral Knee Arthroplasty
MeSH Terms: interventions — Acetaminophen; Orphenadrine; oxycodone-acetaminophen; Hydromorphone; Oxycodone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Control (Active Comparator): Preop acetaminophen IV 1000 mg, Postop oral oxycodone & acetaminophen (5/325 mg) 1 to 2 tabs every 4 hours PRN, and Postop hydromorphone IV 0.5 mg every 4 hours PRN
  Interventions: Drug: Preop acetaminophen IV; Drug: Postop oral oxycodone & acetaminophen; Drug: Postop hydromorphone IV
- Standard (Active Comparator): Preop acetaminophen IV 1000 mg, Preop orphenadrine IV 60 mg, Postop oral orphenadrine 100 mg every 12 hours for 3 doses, Postop oral oxycodone & acetaminophen (5/325 mg) 1 to 2 tabs every 4 hours PRN, Postop hydromorphone IV 0.5 mg every 4 hours PRN
  Interventions: Drug: Preop acetaminophen IV; Drug: Preop orphenadrine IV; Drug: Postop oral oxycodone & acetaminophen; Drug: Postop hydromorphone IV; Drug: Postop oral orphenadrine
- IVAM (Experimental): Preop acetaminophen IV 1000 mg, Preop orphenadrine IV 60 mg, Postop acetaminophen IV 1000 mg every 6 hours for 7 doses, Postop orphenadrine IV 60 mg every 12 hours for 3 doses, Postop oral oxycodone 5 mg 1 to 2 tabs every 4 hours PRN, Postop hydromorphone IV 0.5 mg every 4 hours PRN
  Interventions: Drug: Preop acetaminophen IV; Drug: Preop orphenadrine IV; Drug: Postop hydromorphone IV; Drug: Postop oral oxycodone; Drug: Postop acetaminophen IV; Drug: Postop orphenadrine IV

INTERVENTIONS:
Drug: Preop acetaminophen IV
  Other Names: Ofirmev
Drug: Preop orphenadrine IV
  Other Names: Norflex
  Arms: IVAM; Standard
Drug: Postop oral oxycodone & acetaminophen
  Other Names: Percocet
  Arms: Control; Standard
Drug: Postop hydromorphone IV
  Other Names: Dilaudid
Drug: Postop oral orphenadrine
  Other Names: Norflex
  Arms: Standard
Drug: Postop oral oxycodone
  Other Names: Roxicodone
  Arms: IVAM
Drug: Postop acetaminophen IV
  Other Names: Ofirmev
  Arms: IVAM
Drug: Postop orphenadrine IV
  Other Names: Norflex
  Arms: IVAM

SUMMARY:
This is a prospective, three-arm, randomized, open-label trial to determine if a new pain control protocol which includes regular dosing of intravenous acetaminophen and orphenadrine for 48 hours after total knee surgery reduces the need for opioid pain medication and reduces average pain scores.

DETAILED DESCRIPTION:
This research will be a prospective, three-arm, randomized, open-label trial to assess opioid use and patient reported outcomes after 48 hours of regular IV acetaminophen and muscle relaxant (IVAM) orphenadrine administration following total knee replacement surgery. 180 patients (60 in each arm) will be randomized to receive the standard group treatment, the IVAM group treatment, or to the control grouptreatment.

Standard Group Treatment: includes peripheral nerve single injection or catheter infusions (48 hours) as requested by the surgeon; preoperative (single dose) intravenous acetaminophen (1000 mg) and orphenadrine (60 mg); intraoperative spinal anesthesia or general anesthesia as determined by the anesthesia attending physician; postoperative oral oxycodone (5 mg) with acetaminophen (325 mg) (PRN dosing), oral orphenadrine (100 mg) every 12 hours for 3 doses, and intravenous hydromorphone (PRN dosing) for breakthrough pain.

Control Group Treatment: includes peripheral nerve single injection or catheter infusions (48 hours); preoperative (single dose) intravenous acetaminophen (1000 mg) intraoperative spinal anesthesia or general anesthesia as determined by the anesthesia attending physician; and postoperative oral oxycodone and acetaminophen (PRN dosing), and intravenous hydromorphone (PRN dosing) for breakthrough pain.

IVAM Group Treatment: includes peripheral nerve single injection or catheter infusions (48 hours); preoperative intravenous acetaminophen (1000 mg) and orphenadrine (60 mg); intraoperative spinal anesthesia or general anesthesia as determined by the anesthesia attending physician; postoperative intravenous acetaminophen (1000 mg) every 6 hours routine for total of 8 doses and intravenous orphenadrine (60 mg) every 12 hours for total of 4 doses; oral oxycodone (5 mg) (PRN dosing), and intravenous hydromorphone (PRN dosing) for breakthrough pain.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18-85
2. Primary, unilateral total knee arthroplasty
3. American Society of Anesthesiologist (ASA) physical status I, II, or III

Exclusion Criteria:

1. Chronic pain (as determined by regular opioid use in the month preceding surgery)
2. Preoperative use of centrally acting muscle relaxants in the 24 hours preceding surgery
3. Peripheral regional anesthesia procedures other than femoral nerve injections or catheters for postoperative pain control (such as popliteal block)
4. Severe renal dysfunction, creatinine > 2.0
5. Allergy or other contraindications to use of orphenadrine and/or acetaminophen
6. Pregnant or breast feeding
7. Abnormal Liver Function Tests(LFT) and / or history of chronic/excessive alcohol abuse.
8. History of Hepatitis, B or C,
9. History of cirrhosis or hepatic insufficiency

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 180 (Actual)
Dates: Start 2015-04; Primary Completion 2016-09 (Actual); Study Completion 2016-09 (Actual)

PRIMARY OUTCOMES:
Routine Pain Intensity Scores | 48 hours
  verbal subjective assessment by patient reported to nursing at standard assessment times as an ordinal number between 0 and 10 (inclusive) where 0 is no pain and 10 is the maximum pain imaginable
Abbreviated Pain Intensity Scores | 48 hours
  Verbal subjective assessment by patient reported to nursing at standard assessment times as either "mild", "moderate", or "severe".
Opioid Consumption, | 48 hours
  recorded by nursing with dose and time. Cumulative and total opioid consumption will be analyzed.
Physical therapy metrics/goals | 48 hours
  measured and recorded by physical therapist in daily chart notes quantifying ability to get out of bed, range of motion (in flexion/extension degrees) and average and maximum ambulation (in feet) during postoperative days 0 to 2.

SECONDARY OUTCOMES:
PACU discharge | 48 hours
  Time to discharge from the PACU will be measured from PACU arrival to time of PACU discharge criteria met in minutes.
Hospital Discharge | 48 hours
  Time to discharge from the hospital will be measured from time/date of surgical incision to time/date that hospital discharge criteria is met, measured in hours.
Patient satisfaction | 48 hours
  19 point validated questionnaire of perioperative satisfaction with items for regional anesthesia
Cost as measured by | 48 hours
  study medication acquisition cost reported by pharmacy, study medication administration cost reported by pharmacy and nursing, length of stay cost reported by hospital accounting.

CONTACTS AND LOCATIONS:
Overall Officials: thomas Looke, MD, Principal Investigator — AdventHealth
Locations (1):
- Florida Hospital Winter Park, Winter Park, Florida, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Looke TD, Kluth CT. Effect of preoperative intravenous methocarbamol and intravenous acetaminophen on opioid use after primary total hip and knee replacement. Orthopedics. 2013 Feb;36(2 Suppl):25-32. doi: 10.3928/01477447-20130122-54. PMID 23379573
- [Result] Hidalgo DA, Pusic AL. The role of methocarbamol and intercostal nerve blocks for pain management in breast augmentation. Aesthet Surg J. 2005 Nov-Dec;25(6):571-5. doi: 10.1016/j.asj.2005.09.003. PMID 19338859
- [Result] Schneider MS. Methocarbamol: adjunct therapy for pain management in breast augmentation. Aesthet Surg J. 2002 Jul;22(4):380-1. doi: 10.1067/maj.2002.126750. PMID 19331993
- [Result] Schneider MS. Pain reduction in breast augmentation using methocarbamol. Aesthetic Plast Surg. 1997 Jan-Feb;21(1):23-4. doi: 10.1007/s002669900076. PMID 9204163
- [Result] Gombotz H, Lochner R, Sigl R, Blasl J, Herzer G, Trimmel H. Opiate sparing effect of fixed combination of diclophenac and orphenadrine after unilateral total hip arthroplasty: A double-blind, randomized, placebo-controlled, multi-centre clinical trial. Wien Med Wochenschr. 2010 Nov;160(19-20):526-34. doi: 10.1007/s10354-010-0829-7. Epub 2010 Oct 8. PMID 20890791
- [Result] Malek J, Nedelova I, Lopourova M, Stefan M, Kostal R. [Diclofenac 75mg. and 30 mg. orfenadine (Neodolpasse) versus placebo and piroxicam in postoperative analgesia after arthroscopy]. Acta Chir Orthop Traumatol Cech. 2004;71(2):80-3. Czech. PMID 15151094
- [Result] Sinatra RS, Jahr JS, Reynolds L, Groudine SB, Royal MA, Breitmeyer JB, Viscusi ER. Intravenous acetaminophen for pain after major orthopedic surgery: an expanded analysis. Pain Pract. 2012 Jun;12(5):357-65. doi: 10.1111/j.1533-2500.2011.00514.x. Epub 2011 Oct 19. PMID 22008309
- [Result] Sinatra RS, Jahr JS, Reynolds LW, Viscusi ER, Groudine SB, Payen-Champenois C. Efficacy and safety of single and repeated administration of 1 gram intravenous acetaminophen injection (paracetamol) for pain management after major orthopedic surgery. Anesthesiology. 2005 Apr;102(4):822-31. doi: 10.1097/00000542-200504000-00019. PMID 15791113
- [Result] Korkmaz Dilmen O, Tunali Y, Cakmakkaya OS, Yentur E, Tutuncu AC, Tureci E, Bahar M. Efficacy of intravenous paracetamol, metamizol and lornoxicam on postoperative pain and morphine consumption after lumbar disc surgery. Eur J Anaesthesiol. 2010 May;27(5):428-32. doi: 10.1097/EJA.0b013e32833731a4. PMID 20173643
- [Result] Singla NK, Parulan C, Samson R, Hutchinson J, Bushnell R, Beja EG, Ang R, Royal MA. Plasma and cerebrospinal fluid pharmacokinetic parameters after single-dose administration of intravenous, oral, or rectal acetaminophen. Pain Pract. 2012 Sep;12(7):523-32. doi: 10.1111/j.1533-2500.2012.00556.x. Epub 2012 Apr 24. PMID 22524979
- [Result] Maurice-Szamburski A, Bruder N, Loundou A, Capdevila X, Auquier P. Development and validation of a perioperative satisfaction questionnaire in regional anesthesia. Anesthesiology. 2013 Jan;118(1):78-87. doi: 10.1097/ALN.0b013e31827469f2. PMID 23221859